CLINICAL TRIAL: NCT05850143
Title: EFFECTIVENESS OF SINGLE DOSE ORAL DEXAMETHASONE VERSUS MULTIDOSE PREDNISOLONE FOR TREATMENT OF ACUTE EXACERBATIONS OF ASTHMA AMONG CHILDREN ATTENDING THE EMERGENCY DEPARTMENT OF CHILDREN HOSPITAL, ISLAMABAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: DR. MOHAMMAD ALI ARIF (Other)
Responsible Party: Sponsor-Investigator, DR. MOHAMMAD ALI ARIF, Docter, Shaheed Zulfiqar Ali Bhutto Medical University
Organization: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: ERB/SZABMU/2021-192
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Dexamethasone; Prednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Single dose dexamethsone in acute exacerbation of asthma (Active Comparator)
  Interventions: Drug: Dexamethasone
- Oral Multidose Prednisolone in acute exacerbation of asthma (Active Comparator)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Dexamethasone — Oral Dexamethasone a longer and potent corticosteroid with lesser sideffects and good compliance
  Arms: Oral Single dose dexamethsone in acute exacerbation of asthma
Drug: Prednisolone — Oral Multidose Prednisolone
  Arms: Oral Multidose Prednisolone in acute exacerbation of asthma

SUMMARY:
In this Study i'll compare the effectiveness of two drugs used in acute exacerbation of asthma by their sideffects, complaince and improvement in the PRAM score. The better one would be adapted in our clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* i.Ages 2 to 12years ii. Previous history of asthma as diagnosed by a physician. iii. Presentation with acute exacerbation of asthma with symptoms of cough, wheeze, dyspnoea and oxygen saturation of less than 95% and with PRAM score of more than or equal to 6

Exclusion Criteria:

* i.Critical or life-threatening asthma i.e. patient with silent chest, cyanosis, drowsy, unable to verbalize, marked tachycardia and respiratory distress. ii.Known TB exposure iii.Fever more than 39. 5°C iv.Use of corticosteroids in previous 4 weeks v.Significant co-morbid disease: lung, cardiac, immune, liver, endocrine, neurological or psychiatric

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2019-01-26 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2023-12-26 (Estimated)

PRIMARY OUTCOMES:
Improvement in PRAM score | 4 days
  PRAM will be evaluated at day 4

CONTACTS AND LOCATIONS:
Locations (1):
- Asim Nawaz Niazi, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided